CLINICAL TRIAL: NCT01209637
Title: Impact of Intensive Exercise Training Compared to Inactive Controls on Coronary Collateral Circulation and Plaque Composition in Patients With Significant Stable Coronary Artery Disease
Brief Title: Impact of Intensive Exercise Training on Coronary Collateral Circulation in Patients With Stable CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Sven Möbius-Winkler, PI, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMW 04
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Stable Coronary Artery Disease
Keywords: stable coronary artery disease; significant coronary stenosis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (No Intervention): standard care of coronary artery diseases incl. recommended home based exercise 3x/week
- Exercise training (Active Comparator): exercise training for 4 weeks at 70% of ischemia free individual threshold within a rehabilitation care center
  Interventions: Behavioral: exercise training
- intensive exercise training (Active Comparator): intensive exercise training incl. interval training
  Interventions: Behavioral: Intensive exercise training

INTERVENTIONS:
Behavioral: exercise training — exercise training min. 4 times a day for at least 30 min
  Arms: Exercise training
Behavioral: Intensive exercise training — Intensive exercise training for 4 times / day incl. interval training at 95% individual threshold
  Arms: intensive exercise training

SUMMARY:
Exercise training in patients with coronary artery disease is able to correct several risk factors. Furthermore endothelial function can be improved.

There are some hinds for improved collateral circulation after exercise training, nevertheless there is no study showing significant improvement/ increase in coronary collaterals. This might be due to technique of collateral measurement. Therefore we conduct a study were coronary blod flow before and after 4 weeks of exercise training were measured.

ELIGIBILITY:
Inclusion Criteria:

* stable CAD
* min.1 coronary artery stenosis >50%
* patient is symptomatic ( CCS 1-3)or has documented myocardial ischemia during stress test
* angina threshold >75 Watt
* informed consent

Exclusion Criteria:

* Age <18 oder >75
* akut coronary syndrome within 2 weeks
* LV-EF < 40 %
* significant valve diseases
* reduced patient compliance
* muscular disorder
* bronchial asthma or COLD stadium III and IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
coronary collateral blod flow | 4 weeks

SECONDARY OUTCOMES:
plaque composition within the coronary artery | 4 weeks
  plaque composition measured by virtual histology intravascular ultrasound
MACCE | 4 week, 6 months, 12 months
  major cardiovascular events (death, myocardial infarction, stroke, TIA, coronary revascularisation, hospitalisation)
atherosclerosis parameter within the laboratory | 4 weeks, 3, 6, 12 months
  e.g. wie hs-CRP, HDL, LDL, ges. Cholesterin, Triglyceride, Zytokine, Adipokine, Endocannaboide

CONTACTS AND LOCATIONS:
Overall Officials: Sven Möbius-Winkler, MD, Principal Investigator — Heart Center Leipzig- University Leipzig
Locations (1):
- Heart Center Leipzig- University Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Mobius-Winkler S, Uhlemann M, Adams V, Sandri M, Erbs S, Lenk K, Mangner N, Mueller U, Adam J, Grunze M, Brunner S, Hilberg T, Mende M, Linke AP, Schuler G. Coronary Collateral Growth Induced by Physical Exercise: Results of the Impact of Intensive Exercise Training on Coronary Collateral Circulation in Patients With Stable Coronary Artery Disease (EXCITE) Trial. Circulation. 2016 Apr 12;133(15):1438-48; discussion 1448. doi: 10.1161/CIRCULATIONAHA.115.016442. Epub 2016 Mar 15. PMID 26979085
- [Derived] Uhlemann M, Adams V, Lenk K, Linke A, Erbs S, Adam J, Thiele H, Hilberg T, Gutberlet M, Grunze M, Schuler GC, Mobius-Winkler S. Impact of different exercise training modalities on the coronary collateral circulation and plaque composition in patients with significant coronary artery disease (EXCITE trial): study protocol for a randomized controlled trial. Trials. 2012 Sep 14;13:167. doi: 10.1186/1745-6215-13-167. PMID 22974129